CLINICAL TRIAL: NCT06578702
Title: Evaluation of Intermittent Triple Therapies in Real Life
Acronym: ETRIVIE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9238
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: HIV Infections
Keywords: HIV Infections; Intermittent Triple Therapy
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The strategy of intermittent triple therapy for people living with HIV was validated in France following the randomized clinical trial QUATUOR. There is little data in real life, as shown in the meta-analysis of Parienti JJ et al.

Currently this strategy is proposed by some teams in France, but is not recommended internationally.

The research hypothesis is that intermittent treatment is an effective and safe option in a therapeutic lightening strategy in people living with HIV People living with HIV adults followed in Strasbourg who have benefited from intermittent treatment The expected results will consist of an improvement in knowledge on the efficacy and tolerance of this therapeutic strategy.

ELIGIBILITY:
Inclusion criteria:

* Adult subject (≥ 18 years old)
* Living with HIV monitored at the Trait d'Union/Infectious Diseases department in Strasbourg
* Having benefited from intermittent triple therapy between 01/01/2017 and 31/01/2024

Exclusion criteria:

* Subject (and/or their legal representative if applicable) having expressed their opposition to the reuse of their data for scientific research purposes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subject (≥ 18 years old) living with HIV monitored at the Trait d'Union/Infectious Diseases department in Strasbourg and having benefited from intermittent triple therapy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-02-21 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02-21 (Estimated)

PRIMARY OUTCOMES:
Evaluation of HIV viral load | 48 weeks after reduction of the HIV viral load

CONTACTS AND LOCATIONS:
Locations (1):
- Service Le Trait d'Union - CHU de Strasbourg - France, Strasbourg, France